CLINICAL TRIAL: NCT06415877
Title: The Effect of the Modified Simulation Model on Self-Efficacy, Anxiety, and Academic Motivation in Episiotomy Training
Acronym: Episiotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1111111
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Episiotomy; Anxiety; Simulation
Keywords: episiotomy; anxiety; simulation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): beef tongue stitched
  Interventions: Other: Episio Training
- sham comparator (Sham Comparator): episio model
  Interventions: Other: Episio Training
- experimental group (Experimental): modified tripe coated veal
  Interventions: Other: Episio Training

INTERVENTIONS:
Other: Episio Training — episio repair training

SUMMARY:
It was planned as a randomized controlled study to determine the effect of the modified simulation model on self-efficacy, anxiety and academic motivation in episiotomy training. It will be held online with students from the midwifery department of Osmaniye Korkut Ata University.

ELIGIBILITY:
Inclusion Criteria:

* Midwifery student
* volunteers

Exclusion Criteria:

* involuntary

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
self-efficacy | 1 week
  questionnaire

SECONDARY OUTCOMES:
academic motivation | 1 week
  questionnaire